CLINICAL TRIAL: NCT05289258
Title: Effectiveness of Cognitive Rehabilitation and the Unified Barlow Protocol (UP) in Cancer Survivors for Cognitive Impairments: a Randomized Controlled Trial
Brief Title: Unified Barlow Protocol (UP) in Cancer Survivors for Cognitive Impairments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Córdoba (Other)
Responsible Party: Principal Investigator, Francisco Garcia Torres, Principal Investigator, Universidad de Córdoba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1380800-R
Record Dates: First submitted 2021-12-28; First posted 2022-03-21 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Cancer, Breast
Keywords: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP); cognitive impairments; quality of life; anxiety and depression.
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This study is a three-arm randomized clinical trial, with a pre-post-follow-up repeated measures intergroup design.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Neuropsychological treatment (Active Comparator): Combination of different neuropsychological rehabilitation programs
  Interventions: Behavioral: Neuropsychological treatment
- Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (PU). (Experimental): This intervention focuses on a deficit in emotional regulation common in all emotional disorders (ED).
  Interventions: Behavioral: Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (PU).
- Waitlist group (Other): The control group will receive the Adapted Mnesic Cognitive Training (ACTIVE) (Jobe, et al., 2001), as well as the Insight (Posit Science) program (Mahncke et al., 2006) once the interventions in groups 1 and 2 have been completed.
  Interventions: Behavioral: Waitlist group

INTERVENTIONS:
Behavioral: Neuropsychological treatment — combination of the programs tested by (Von Ah et al. 2012). These programs are, on the one hand, a cognitive training adapted from the Advanced Cognitive Training for Independent and Vital Elderly (ACTIVE) (Jobe et al., 2001) and, on the other, a processing speed training using the Insight program (from Posit Science) (Mahncke et al., 2006). The first consists of teaching patients memorization techniques, and the second consists of a series of exercises on information processing of varying difficulty. These exercises automatically adjust your difficulty to maintain an 85% rate of return. Treatment is carried out in groups of 10 cancer survivors. It consists of 10 weekly sessions of 2 hours each (the first hour for memory training and the second for processing speed exercises). In order to improve the adherence to treatment of the participants, emails and telephone text messages will be sent with reminders of appointments and tasks to be performed.
  Arms: Neuropsychological treatment
Behavioral: Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (PU). — This intervention focuses on a deficit in emotional regulation common in all emotional disorders (ED). Therefore, it focuses on the adaptive value of emotions and promotes tolerance to intense emotions as well as the identification and modification of dysfunctional emotional regulation strategies. Patients receive 10 group therapy sessions (3-5 cancer survivors per group) with all PU modules (Barlow et al., 2011). The Spanish version of the therapist's guide and the patient's workbook are used (Barlow et al., 2015). All patients receive the workbook to help them read the contents of each session, do the recommended exercises between sessions, and to help them once the treatment is finished. The treatment lasts 10 weeks (one session a week). As in the previous intervention group, emails and telephone text messages will be used with reminders of appointments and tasks to be carried out.
  Arms: Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (PU).
Behavioral: Waitlist group — The control group will receive the Adapted Mnesic Cognitive Training (ACTIVE) (Jobe, et al., 2001), as well as the Insight (Posit Science) program (Mahncke et al., 2006) once the interventions in groups 1 and 2 have been completed.
  Arms: Waitlist group

SUMMARY:
Background: Cognitive impairment appears frequently in cancer survivors, negatively affecting the quality of life and emotional well-being of patients. This study compares the effectiveness of a well-established treatment (cognitive rehabilitation) with the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP) to alleviate these cognitive deficits and evaluate its effect on anxiety-depressive symptoms and the quality of life of survivors.

Methods: A three-arm randomized superiority clinical trial, with a pre-post and follow-up repeated measures and intergroup design with a 1:1:1 allocation ratio will be carried out. A hundred and twenty-three breast cancer survivors with mild to moderate cognitive impairment will be randomly assigned to one of the interventions of the study: cognitive rehabilitation intervention group, an intervention group with UP intervention, or a control group on the waiting list. The primary outcome is to observe a significant improvement in cognitive function and quality of life in both intervention groups and a significant decrease in emotional impairments in comparison with the waitlist group. These results will be maintained at six months of follow-up.

Discussion: The aim of this work is to test the efficacy of the Unified Barlow Protocol in reducing cognitive deficits in breast cancer survivors. The results of this trial may be useful in reducing the presence of cognitive problems in survivors and improving their emotional state and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Cancer diagnosis, stages I-III.
* Cancer type: Breast.
* Have received the last chemotherapy session in the last 6 months and a maximum of 6 years of treatment completion.
* Probable or mild to moderate cognitive impairment (score between 26 and 10 points according to the MMSE).
* Ability to be fluent in Spanish.
* Not currently participating in another clinical trial.
* Not currently receiving other psychological treatment

Exclusion Criteria:

* Men and women aged > 70 years.
* Diagnosis of cancer, stage IV or other types of cancer.
* Last chemotherapy session < 6 months or > 6 years.
* No cognitive impairment (MMSE score between 30 and 27 points).
* Diagnosis of mental disorder (including substance abuse) prior to cancer diagnosis.
* Relapse in disease after chemotherapy treatment is completed.
* Neurodevelopmental Disorder Diagnosis.
* Diagnosis of diseases that affect cognitive performance such as: hypertension, cardiac diseases, epilepsy, dementias, multiple sclerosis, functional disorders (fibromyalgia, chronic fatigue syndrome, irritable bowel syndrome, post-concussion syndrome, whiplash syndrome), CNS infections (HIV, encephalitis), metabolic disorders (diabetes, B12 deficiency), obstructive sleep apnea, brain damage (stroke, TBI, CNS cancer) and use of medications / substances that interfere with cognitive function such as pregabalin, gabapentin, topiramate, antidepressants tricyclics, sodium valproate, anticholinergics, methylphenidate, typical antipsychotics.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional assessment of Cancer Therapy-Cognitive Function, version 3. (FACT-Cog). | Change of mean scores from baseline to immediately after intervention
  This is an instrument developed to assess chemotherapy-induced cognitive problems in cancer patients. It includes four different subscales: Perceived Cognitive Impairments (score range from 0-72), Impact of Perceived Cognitive Impairments on QoL (score range from 0-16), Comments from Others (score range from 0-16), and Perceived Cognitive Abilities (scores range from 0-28) that are scored using a Likert scale of five points from 0 (never) to 4 (several times a day). The higher the score, the better the cognitive function
Memory Failures Everyday (MFE-30). | Change of mean scores from baseline to immediately after intervention
  It is a unifactorial questionnaire that measures a single construct: "cognitive complaints". It is made up of 30 items that are answered on a 5-point Likert scale from 1 (never) to 4 (always or almost always) with higher scores indicate poorer memory function. Scores are from 1 to with higher scores indicating higher memory impairments
Hopkins Verbal Learning Test-Revised (HVLT-R). | Change of mean scores from baseline to immediately after intervention
  This test measures primary and secondary memory, the rate of verbal learning throughout three trials, as well as three forms of mnesic organization: serial ordering, semantic grouping, and subjective organization. The test consists of a list of 12 words that are presented orally at a speed of one word for every two seconds. a higher number of words is interpreted as better recall and recognition
Trail Making Test (TMT). | Change of mean scores from baseline to immediately after intervention
  The TMT consists of two parts: Part A measures attention, processing speed, visual search, and working memory; on the other hand, part B is used to measure attention, executive function (cognitive flexibility, ability to change tasks, coordination of categories), working memory, visual-motor skills and processing speed. A greater time to complete the tasks is interpreted as a greater deterioration
Controlled Oral Word Association Test (COWAT). | Change of mean scores from baseline to immediately after intervention
  The COWAT is a test that measures verbal fluency and is a recognized and sensitive indicator of cognitive functioning. the participant has to say as many words as possible in one minute, and a greater number of words is associated with greater verbal fluency.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Change of mean scores from baseline to immediately after intervention]
  This scale is used to assess anxiety and depression in a hospital settings. It is made up of 14 items (7 for anxiety and 7 for depression), which are answered on a scale from 0 to 3, with maximum values of 21 in each of the subscales. Higher scores indicates the presence of anxiety and depression.
Quality of Life scores using EORTC QLQ C-30. | Change of mean scores from baseline to immediately after intervention]
  EORTC QLQ C-30 (version 3), this is an instrument developed to assess the quality of life in cancer patients using 30 questions that refer to the quality of life experienced by the patient during the last week. The first twenty-eight items include questions about different symptoms and are answered on a scale that ranges from 1 (not at all) to 4 (a lot), while the last two ask patients about the perception of their global health and quality of life in a scale from 1 (terrible) to 7 (excellent). The different items are grouped into functional scales (physical / role / emotional / cognitive / social and global) and symptom scale (fatigue / nausea and vomiting / dyspnea / sleep problems / loss of appetite / constipation / diarrhea and financial impact ). Higher scores indicates a better function.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Reina Sofía University Hospital, Córdoba, Córdoba

IPD SHARING:
Plan to Share IPD: No
not applicable for this trial

REFERENCES:
- [Derived] Garcia-Torres F, Tejero-Perea A, Gomez-Solis A, Castillo-Mayen R, Jaen-Moreno MJ, Luque B, Galvez-Lara M, Sanchez-Raya A, Jablonski M, Rodriguez-Alonso B, Aranda E. Effectiveness of the Unified Barlow Protocol (UP) and neuropsychological treatment in cancer survivors for cognitive impairments: study protocol for a randomized controlled trial. Trials. 2022 Sep 30;23(1):819. doi: 10.1186/s13063-022-06731-w. PMID 36175973